CLINICAL TRIAL: NCT06700824
Title: MATRISS-II. Matrix Therapy to Reduce Ischemic Stroke Sequelae-II. a Randomized-double Blinded- Placebo Controlled Trial to Assess the Efficacy and Safety of OTR4132-MD in Patients with Acute Ischemic Stroke
Brief Title: A Trial to Assess the Efficacy and Safety of OTR4132-MD in Patients with Acute Ischemic Stroke
Acronym: MATRISS-II
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Organ, Tissue, Regeneration, Repair and Replacement (Industry)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MATRISS-II; 2024-A01526-41 (Other: IDRCB)
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Endovascular Thrombectomy; Ischemic Cerebrovascular Accident
Keywords: OTR4132; RGTA; neuroprotective agents; randomized controlled trial; ischemic stroke; endovacular thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OTR4132 (Experimental): OTR4132 is a new ReGeneraTing Agent (RGTA®) which is a polymer of glucose (α-1,6 bounds, i.e. dextran backbone) engineered to mimic heparan sulphate (HS) in all three mechanical functions (extracellular matrix scaffold element, protector of matrix pro-teins and cellular communication peptides storage sites) but differ from HS by their resistance to glycanases. OTR4132 allows a restoration of the matrix architecture which secondarily facilitates cell survival and recovery at the site of injury.
  Interventions: Device: OTR4132
- Placebo (Placebo Comparator): Saline solution
  Interventions: Device: Placebo

INTERVENTIONS:
Device: OTR4132 — OTR4132 is a new ReGeneraTing Agent (RGTA®) which is a polymer of glucose (α-1,6 bounds, i.e. dextran backbone) engineered to mimic heparan sulphate (HS) in all three mechanical functions (extracellular matrix scaffold element, protector of matrix pro-teins and cellular communication peptides storage sites) but differ from HS by their resistance to glycanases. OTR4132 allows a restoration of the matrix architecture which secondarily facilitates cell survival and recovery at the site of injury.
  Arms: OTR4132
Device: Placebo — saline solution
  Arms: Placebo

SUMMARY:
The MaTRISS 2 study is a phase 2 randomized, double-blinded and placebo-controlled trial aimed at recruiting 60 subjects (30 placebo and 30 active) from 15 stroke centers in France. The main objective will be to assess the efficacy of OTR4132-MD in patients with anterior ischemic stroke after endovascular thrombectomy. One dose will be tested (2 mg) against placebo. The main outcomes will be NIHSS (neurological score) at 24 hours, rate of intracranial hemorrhages at 24 hours, MRI lesion volume at 3 months and neurological scores at 3 months.

DETAILED DESCRIPTION:
* The aim of the study is to confirm previous safety and encouraging efficacy data obtained from the MATRISS first-in man study and animal studies.

  . This is a prospective double-blinded placebo-controlled trial. The trial will recruit 60 subjects (30 per group) with anterior circulation acute ischemic stroke (AIS) re-vascularized (TICI score 2b - 3) by endovascular thrombectomy. Subjects will be followed for 3 months after a single administration of OTR4132-MD or placebo.
* The study is double blinded and there is no way to distinguish the active product from the placebo. Neither the treating nor evaluating physicians, nor the patients, will be informed of the allocation of the treatment before database lock and the end of the trial.
* The use of a placebo is justified by the absence of any neuroprotector approved in France in this indication so there is no comparator. The administration of OTR4132-MD or Placebo will be done in addition to the best standard of care and does not result in any additional po-tentially harmful procedure.
* The study will include 60 patients (30 in the active group and 30 in the placebo group) which is considered sufficient to demonstrate superiority of treatment over placebo with a 5% risk two-sided level (see sample size calculation).
* The study will evaluate a single dose of OTR4132-MD (2 mg) over Placebo. This dose has been selected as the highest and safest dose tested in the previous MATRISS dose-escalation study.
* A 3 months-follow-up period is estimated sufficient to evaluate the residual disability and is recommended in the guideline "Points to consider on clinical investigation of medicinal products for the treatment of acute stroke" (EMA, 2001, CPMP/EWP/560/98).
* A Data Safety Monitoring Board (DSMB) will be set up. It will consist of three medical experts in neurology and stroke trials. Other relevant expertise will be consulted if deemed neces-sary. The members of the committee will review interim blinded safety and efficacy study da-ta. Unblinding procedures will be set up in individual cases if deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85 years
2. Acute ischemic stroke in anterior circulation territory, identified by magnetic resonance imaging (MRI).
3. Occlusion of anterior circulation i.e. carotid artery (ICA) or proximal middle cerebral artery (MCA) (M1 and/or M2 segment)
4. Endovascular thrombectomy (with or without previous intravenous thrombolysis)
5. Recanalization confirmed by angiography after endovascular treatment: TICI grade 2b - 3
6. NIHSS (National Institute of Health Stroke Scale/Score) ≥ 11
7. Pre-stroke modified Rankin Score (mRS): 0 or 1
8. Patient* or legally authorized representative (family member or trusted person if patient unable to give consent) or independent physician (if patient unable to give consent and if an authorized representative cannot be reached) has signed informed consent.

   * Patients unable to give consent at baseline will go through a deferred consent procedure to continue the study

Exclusion Criteria:

1. Previous symptomatic stroke with permanent sequelae
2. Pre-existing medical, neurological, or psychiatric disease that would confound the neurological evaluation
3. Contraindication to MRI
4. Stroke lesion not visible on MRI
5. History of allergy or anaphylactic reactions to any of the ingredients of OTR4132-MD or heparinoids
6. History of hypersensitivity or anaphylactic reactions to iodinated contrast media
7. Intracranial tumor at inclusion
8. Pregnant or breastfeeding women
9. Severe renal failure with glomerular filtration rate (GFR) < 30 mL/min
10. Severe uncontrolled arterial hypertension e.g. systolic blood pressure > 185 mmHg or diastolic blood pressure > 110 mmHg, or intravenous medication necessary to reduce blood pressure
11. Life expectancy of less than 3 months or co-morbidities that could influence the study results or would complicate assessment of outcomes (e.g. dementia, psychiatric disease) or would make clinical follow-up difficult
12. Increased risk of hemorrhage (for instance medical history of significant bleeding disorders, major surgery or significant trauma in the past 3 months, any history of suspected intracranial hemorrhage, symptoms suggestive of subarachnoid hemorrhage, even if the MRI is normal, international normalized ratio (INR)>1.3 or activated partial thromboplastin time (aPTT)>ULN (upper limit of normal)
13. Suspected cerebral vasculitis based on medical history and imaging
14. Occlusions in multiple vascular territories
15. Evidence of any prior intracranial intervention (i.e. neurosurgery, endovascular intervention)
16. Worsening of medical or neurological conditions or per-procedures complications
17. Any other serious, advanced, or terminal illness (investigator judgment)
18. Current participation in another therapeutic investigation (drug or device)
19. The patient is not a member or beneficiary of the French social security system

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Baseline-Adjusted 24-Hour NIHSS | 24 hours
  The NIH Stroke Scale (NIHSS) is based on the collection of 15 clinical neurological items. It allows for an accurate and rapid assessment of observed deficits. A large number of publications have shown that the NIHSS score at 24 hours is the best prognostic factor for long-term functional disability and is closely correlated with disability scores at 3 months. An NIHSS score between 1 and 4 means a minor stroke, between 5 and 15, a moderate stroke, above 15 points, a severe stroke. The maximum score is 42

SECONDARY OUTCOMES:
Change in modified Rankin scale (mRS) at 3 months | 3 months
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire. The Modified Rankin Score (mRS) is the most widely used outcome measure in stroke clinical trials. Standardized interviews to obtain a mRS score are recommended at 3 months (90 days) following hospital discharge. The mRS will be used as a continuous endpoint (change in mRS at 3 months and in a responder analysis (mRS 0-2 at 3 months).
Changes in total lesion volume from baseline to 3 months (MRI) | 3 months
  Follow-up infarct volume is a more direct measure of biological effect of treatment. Infarct volume is less likely to be confounded by intervening comorbid illness, rehabilitation therapy, or non-stroke related pathology.
  volumetric analyses will be analyzed by an independent core laboratory
The rate of Intracranial hemorrhage at 24-hour | 24 hours
  The rate of Intracranial hemorrhage at 24-hour based on Heidelberg classification is considered an important endpoint to assess the potential performance of OTR4132-MD in the repair of the blood brain barrier
Barthel Index at 3-months | 3 months
  Modified Barthel Index (from 0 to 20) is a measure of physical disability used widely to assess behaviour relating to activities of daily living. It measures what patients do in practice. Assessment is made by anyone who knows the patient well.
  100: normal <99 represents slight dependency <90 represents moderate disability <60 represents severe disability >20 represents total dependency

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Detante, MD, Principal Investigator — Centre Hospitalier Universitaire Grenoble Alpes
Locations (15):
- France (15):
  - Centre Hospitalier Universi-taire de Bordeaux-Hôpital Pellegrin, Bordeaux
  - Centre hospitalier universi-taire de Brest (Cavale Blanche), Brest
  - CHU Henri-Mondor, Créteil
  - Centre Hospitalier Universitaire de Martinique, Fort de France
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - Centre Hospitalier Régional Universitaire de Lille- Hôpital Roger Salengro, Lille
  - Hôpitaux Universitaires De Marseille Timone-AP-HM, Marseille
  - Centre Hospitalier Régional Universitaire de Nancy, Nancy
  - UIC Imagerie et Neurovasculaire CHU de Nantes, Nantes
  - Hôpital de la Pitié Salpêtrière - AP-HP, Paris
  - Hôpital Fondation Adolphe de Rothschild Service de neuro-vasculaire, Paris
  - GHU Paris Psychiatrie & Neurosciences, Paris
  - Centre Hospitalier Universitaire de la Guadeloupe, Pointe à Pitre
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: Undecided